CLINICAL TRIAL: NCT06407063
Title: Long-term Frequency of Reoperations After Micro-decompression Alone Versus Decompression and Instrumented Fusion in Patients With Lumbar Spinal Stenosis and Degenerative Spondylolisthesis
Brief Title: Long-term Reoperations After Lumbar Spinal Stenosis Surgery
Status: Recruiting | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other); Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2813
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Degenerative Lumbar Spondylolisthesis
Keywords: Degenerative Spondylolisthesis; Treatment; Decompression alone; Instrumented fusion; Reoperations
MeSH Terms: interventions — Decompression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated for Degenerative Spondylolisthesis: Patients operated for Degenerative Spondylolisthesis with Lumbar Spinal Stenosis
  Interventions: Procedure: Micro-decompression alone; Procedure: Decompression and instrumented fusion

INTERVENTIONS:
Procedure: Micro-decompression alone — In surgical treatment of Degenerative Spondylolisthesis patients are operated on with a midline-preserving decompression without fusion
Procedure: Decompression and instrumented fusion — In surgical treatment of Degenerative Spondylolisthesis patients are operated on with a decompression followed by an instrumental fusion with or without an additional cage

SUMMARY:
Severe and persisting pain and disability due to a degenerative narrowing of the spinal canal, lumbar spinal stenosis, can be operated with a simple surgical decompression. Sometimes, there is also a slippage of vertebra, degenerative spondylolisthesis. In such cases, instrumental stabilization (e.g. screws and rods) has been recommended. Even though additional fusion is more complex and riskier, and evidence in high-quality Scandinavian studies shows that it is unnecessary, decompression plus fusion is still the treatment of choice in the USA and most European countries. This reluctance to change clinical practice is mainly due to concerns about long-term results, especially higher reoperation rates among patients operated with decompression only. This register-based non-inferiority study aims to assess long-term reoperations among those treated with and without additional fusion surgery.

DETAILED DESCRIPTION:
The use of fusion surgery in addition to decompression in the treatment of degenerative lumbar spondylolisthesis (DS) with spinal stenosis (LSS) is a long-standing controversy in spine surgery. The main goal of LSS surgery is to decompress the nerve roots. In the 1990s, two observational studies recommended that decompression with additional fusion should be the treatment of choice. Consequently, the practice shifted towards more complex fusion procedures. In 2016, Swedish and one American randomized controlled trials (RCTs), one Swedish and one American, reported conflicting data about reoperations. The study from the US showed a higher frequency of reoperations after decompression only compared to the decompression and fusion, while the Swedish study showed no difference. In 2020, Austevoll et. al. published a study from the Norwegian registry for spine surgery (NORspine) comparing relative effectiveness micro-decompression alone vs decompression and instrumented fusion (5). This study had a non-inferiority design, similar to the RCT published by the same author in 2021 (6). Both studies concluded that micro-decompression alone was non-inferior to decompression and instrumented fusion regarding clinical outcomes and reoperation rates. Despite an increasing number of studies showing no extra benefits from the more risky and complex additional fusion procedures, the surgical practice has changed little outside Scandinavia. This is probably due to the concerns about subsequent instability and higher long-term reoperation rates among those operated with decompression only.

This study is a long-term follow-up of the NORspine relative effectiveness study from 2020, comprising 794 patients having an index operation for LSS and DS between September 19th 2007 and December 21st 2015 (index study). The present study aims to assess long-term reoperations resulting from everyday clinical practice. The investigators alternative hypothesis is that micro-decompression alone is non-inferior to decompression plus instrumented fusion. The non-inferior margin is specified to correspond to a number needed to treat = 8 to avoid reoperation on one patient in the first 10 postoperative years, corresponding to a between-group difference of 12.5 percentage points (100/8 = 12.5).

The dataset will contain NORspine data at baseline, 3 months, one year and long-term follow-up performed at 7 to 15 years (NCT03469791). NORspine also provides dates of death for all deceased patients. The Norwegian Patient Registry (NPR) will serve as an external data source, providing data about all reoperations until August 31st 2023 and the baseline Charlson Comorbidity Index (CCI). NPR data will ensure follow-up of 8 to 16 years concerning reoperations. For these cases, a review the electronic health records to validate NPR data regarding classification of reoperation (level, indication, surgical technique, total number of reoperations, spinal cord stimulation, reoperations within 90 days after the index operation, participation in other studies).

In the index study propensity score matching (PSM) was performed to reduce the risk of selection bias due to case-mix. The same PSM will be used in the present study. matching. The following parameters were included in the calculation of the propensity score: Age; Gender; American Society of Anaesthesiologists (ASA) grade; Body Mass Index (BMI); Smoking, Oswestry Disability Index (ODI), Numeric Rating Scale for leg pain and back pain, Euroqol 5D (EQ-5D-3L), foraminal stenosis, degenerative disc disease, predominating back pain, number of levels operated on and neurological palsy. The propensity scores were derived from a logistic regression model and reflected a patient's theoretical baseline probability for being instrumentally fused. Using the '1:1 matching without replacement' method, pairs of fused and non-fused patients with a difference in propensity scores less than 0.2 in the logit of the standard deviation were formed. Statistical Package for the Social Sciences (SPSS) version 24 was used for propensity score matching. For comparison, complete case analyses will also be performed.

In this non-inferiority designed study, the primary outcome will be the occurrence of a reoperation, defined as new lumbar spine operation more than 90 days after the index operation until August 31st 2023 (range: from 8 to 16 years after the primary operation. The rate of reoperation within 90 days (n%) of will be reported separately, and will be classified as a complication to the index operation. Survival analysis will be used to detect whether the probability for reoperation during the first 10 years is more than 12.5 % higher (non-inferiority margin) in the micro-decompression group than in the decompression and instrumented fusion group or not. This is to be tested by deriving a 90 % confidence interval (CI) for the difference of the survival function (S(t)) at 10 years between the groups (S(t) in decompression and instrumented fusion group - S(t) in micro-decompression group) where t = 10 years. Thus, a lower limit of the CI above -0.125 will indicate that, in an everyday clinical practice setting, micro-decompression would be non-inferior to decompression and instrumented fusion regarding the risk of reoperation. In addition, the investigators will report survival functions and observed reoperation rates at multiple timepoints (2, 5 and 10 years), hazard ratio (HR) for reoperation (at 2, 5 and 10 years, as well as complications (including reoperations within 90 days). The indication for reoperation, surgical techniques and risk factors associated with reoperation will also be investigated.

For the power analysis conducted with PASS 2019, two assumptions were made. 1) Expected reoperation rate: Based on NORspine data, about 27.1 % of lumbar surgical procedures are performed on patients previously operated. Using this as a proxy for the expected probability of reoperation in the total cohort. 2) HR = 1.6 (decompression and instrumented fusion) approximates the event ratio between the groups. Applying these assumptions, choosing a type 1 error = 0.05 and power 0.8 gives sample size = 269 per group. The index study had a sample size of 285 in each PSM group. Since the present study will use national administrative registries and patient's health records, substantial loss to follow-up is not expected.

For statistical analyses SAS Enterprise Guide 8.3 will be used, including descriptive statistics, tests for data distribution, cross-tabulations with χ2 test, Student t-tests, and Mann-Whitney U tests. Reoperation survival, hazard and rates will be assessed by stratified log-rank test, cox regression modelling (time-dependent if the proportional hazard assumption is violated), Kaplan-Meier plots and multivariable regression analyses.

ELIGIBILITY:
Inclusion Criteria:

* operated between September 2007 and December 2015 labeled in the registry with both 'Spinal stenosis' and 'Degenerative spondylolisthesis'
* operated on with decompression with or without an additional fusion

Exclusion Criteria:

* operated with an anterior approach
* had a former operation at index Level
* was labeled with a degenerative scoliosis
* was operated in more than 2 Levels
* was operated with non-instrumented fusion
* operated with a standard laminectomy with removing of the posterior midline structures or operated without magnifying devices was excluded from the micro-decompression group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is defined by the NORspine registry and contains all patients in the register in the priode September 19 2007 to Desember 21 2015 that fulfil the eligibility criteria. The NORspine register cases in a specialiced health care setting from the Norwegian providers of lumbar spine surgery.
Sampling Method: Probability Sample
Enrollment: 794 (Estimated)
Dates: Start 2007-09-19 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Estimated reoperations rate (n, %) at 10 years follow-up (Survival function (S(t), t=10 years) for first reoperation) by treatment group | From date of index operation (2007-2015) until end of follow up August 31st 2023
  Survival function for a reoperation at 10 years. A new operation in the lumbosacral spine (excluding surgery for tumor and trauma) during follow up, occurring more than 90 days after index surgery is defined as reoperation.

SECONDARY OUTCOMES:
Hazard ratio(s) and survival functions for reoperation and reoperations rates by treatment group. | From date of index operation (2007-2015) until end of follow up August 31st 2023
  Hazard ratio(s) and survival functions for reoperation and reoperations rates, reported at 2, 5 and 10 years follow-up. A new operation in the lumbosacral spine (excluding surgery for tumor and trauma) during follow up, occurring more than 90 days after index surgery is defined as reoperation.
Rate of reoperations within 90 days after index surgery (n %) by treatment group. | From date of index operation (2007-2015) until 90 days after index surgery
  This is reported separately since early reoperations (within 90 days) are categorized as complications in the NORspine (n %)
Other complications (n %) by treatment group | Reported at baseline and 3 months after the index operation
  Complications (n %) related to index operation reported in NORspine. Surgeon and patient reported. e.g dural tear, postoperative haematoma, surgical site infection, thromboembolism (DVT, LE), pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Tore Solberg, Prof, Principal Investigator — University Hospital of North Norway
Locations (1):
- University hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No
No sharing is planed due to the sensitive nature of the research data

REFERENCES:
- [Background] Herkowitz HN, Kurz LT. Degenerative lumbar spondylolisthesis with spinal stenosis. A prospective study comparing decompression with decompression and intertransverse process arthrodesis. J Bone Joint Surg Am. 1991 Jul;73(6):802-8. PMID 2071615
- [Background] Bridwell KH, Sedgewick TA, O'Brien MF, Lenke LG, Baldus C. The role of fusion and instrumentation in the treatment of degenerative spondylolisthesis with spinal stenosis. J Spinal Disord. 1993 Dec;6(6):461-72. doi: 10.1097/00002517-199306060-00001. PMID 8130395
- [Background] Forsth P, Olafsson G, Carlsson T, Frost A, Borgstrom F, Fritzell P, Ohagen P, Michaelsson K, Sanden B. A Randomized, Controlled Trial of Fusion Surgery for Lumbar Spinal Stenosis. N Engl J Med. 2016 Apr 14;374(15):1413-23. doi: 10.1056/NEJMoa1513721. PMID 27074066
- [Background] Ghogawala Z, Dziura J, Butler WE, Dai F, Terrin N, Magge SN, Coumans JV, Harrington JF, Amin-Hanjani S, Schwartz JS, Sonntag VK, Barker FG 2nd, Benzel EC. Laminectomy plus Fusion versus Laminectomy Alone for Lumbar Spondylolisthesis. N Engl J Med. 2016 Apr 14;374(15):1424-34. doi: 10.1056/NEJMoa1508788. PMID 27074067
- [Background] Austevoll IM, Gjestad R, Solberg T, Storheim K, Brox JI, Hermansen E, Rekeland F, Indrekvam K, Hellum C. Comparative Effectiveness of Microdecompression Alone vs Decompression Plus Instrumented Fusion in Lumbar Degenerative Spondylolisthesis. JAMA Netw Open. 2020 Sep 1;3(9):e2015015. doi: 10.1001/jamanetworkopen.2020.15015. PMID 32910195
- [Background] Austevoll IM, Hermansen E, Fagerland MW, Storheim K, Brox JI, Solberg T, Rekeland F, Franssen E, Weber C, Brisby H, Grundnes O, Algaard KRH, Boker T, Banitalebi H, Indrekvam K, Hellum C; NORDSTEN-DS Investigators. Decompression with or without Fusion in Degenerative Lumbar Spondylolisthesis. N Engl J Med. 2021 Aug 5;385(6):526-538. doi: 10.1056/NEJMoa2100990. PMID 34347953